CLINICAL TRIAL: NCT05734209
Title: How Does Eating Behavior and Hunger in Virtual Reality Meals Compare to Real Meals? A Randomized Crossover Study
Brief Title: How Does Eating Behavior and Hunger in Virtual Reality Meals Compare to Real Meals?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Billy Langlet, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-04249
Record Dates: First submitted 2022-12-15; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Hunger

STUDY DESIGN:
Intervention Model Description: Randomized crossover study with 2 repeats. Each person participated in two virtual meals and two real meals in random order.
Masking Description: Masking was not possible in the current study, since it was obvious if you were eating virtual or real food. However, participants were not aware of the aim of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual, then real meal (Experimental): Participant first had two lunch sessions eating virtual food (meal), with a wash-out period of three days. Participants then had two lunch sessions eating real food (meal), with a wash-out period of three days.
  Interventions: Behavioral: Virtual food; Behavioral: Real food
- Real, then virtual meal (Experimental): Participant first had two lunch sessions eating real food (meal), with a wash-out period of three days. Participants then had two lunch sessions eating virtual food (meal), with a wash-out period of three days.
  Interventions: Behavioral: Virtual food; Behavioral: Real food

INTERVENTIONS:
Behavioral: Virtual food — Virtual food eaten using immersive virtual reality equipment
Behavioral: Real food — Real food eaten using regular utensils

SUMMARY:
Objective: To investigate the differences between eating virtual and real-life meals and test the hypothesis that eating a virtual meal can reduce hunger among healthy women.

Methods: Twenty healthy women will be recruited and partake in a randomized crossover study. The subjects will be asked to eat one introduction meal, two real meals, and two virtual meals, all containing real or virtual meatballs and potatoes. The real meals will be eaten on a plate placed on a scale which communicates with analytical software on a computer. The virtual meals will be eaten in a room, where participants are seated on a real chair in front of a real table, and fitted with the virtual-reality equipment. The eating behavior for both the real and virtual meals will be filmed. Hunger will be measured before and after the meals using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 kg/m2 to 29 kg/m2
* "normal" physical activity (measured using the short version of the international physical activity questionnaire, IPAQ)

Exclusion Criteria:

* pregnant or breastfeeding
* smoker
* temporomandibular disorder
* recent serious dental surgery (last 6 months)
* undergoing treatments known to affect appetite (e.g., use of some psychotropic drugs)
* previous history of eating disorders
* vegetarian
* aversion to the food served

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-03 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Difference in hunger before to after meal | Before to after meal (on average around 10 minutes)
  Rated on visual analogue scale (range 0 - 100)

SECONDARY OUTCOMES:
Food intake | During meal (around 10 minutes)
  Grams of food ingested
Meal duration | During meal (around 10 minutes)
  Minute duration of the meal
Forkfuls | During meal (around 10 minutes)
  Number of times participant took food from the plate
Additions | During meal (around 10 minutes)
  Number of times the participant added food to the plate
Chews | During meal (around 10 minutes)
  Number of times the participant chewed the food

CONTACTS AND LOCATIONS:
Overall Officials: Billy S Langlet, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Huddinge, Sweden

REFERENCES:
- [Derived] Glympi A, Odegi D, Zandian M, Sodersten P, Bergh C, Langlet B. Eating Behavior and Satiety With Virtual Reality Meals Compared With Real Meals: Randomized Crossover Study. JMIR Serious Games. 2023 Aug 10;11:e44348. doi: 10.2196/44348. PMID 37561558